CLINICAL TRIAL: NCT06551727
Title: Antithrombotic Therapy With Regulation of Blood Pressure in Non-Cardioembolic Progressive Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, LI LONGXUAN, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024213
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): After stroke progression, all patients receive dual antiplatelet therapy (aspirin 100mg/day combined with clopidogrel 75mg/day) for the first 21 days, except in cases of cerebral hemorrhage. After this period, they continue to take aspirin 100mg/day orally for the long term.
  Interventions: Other: Control group
- Intervention group (Experimental): After stroke progression, all patients receive dual antiplatelet therapy (aspirin 100mg/day combined with clopidogrel 75mg/day) for the first 21 days, except in cases of cerebral hemorrhage. After this period, they continue to take aspirin 100mg/day orally for the long term. In terms of blood pressure control, medications such as dopamine, metaraminol, or midodrine are used to achieve a systolic blood pressure target range of 160-180 mmHg within 1 h of random assignment and to maintain this target for 7 days (or death, should this event occur earlier). BP measurements are routinely captured using automated devices fitted to the unaffected arm, following the protocol recommended by the standard guideline. The readings are taken at 15-minute intervals for the initial hour, hourly from the first to the sixth hour, every six hours from 6 to 24 hours, and then twice daily for 7 days (or death, if earlier). Subsequently, these data are uploaded into the research database.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — After stroke progression, all patients receive dual antiplatelet therapy (aspirin 100mg/day combined with clopidogrel 75mg/day) for the first 21 days, except in cases of cerebral hemorrhage. After this period, they continue to take aspirin 100mg/day orally for the long term.
  In terms of blood pressure control, medications such as dopamine, metaraminol, or midodrine are used to achieve a systolic blood pressure target range of 160-180 mmHg within 1 h of random assignment and to maintain this target for 7 days (or death, should this event occur earlier). BP measurements are routinely captured using automated devices fitted to the unaffected arm, following the protocol recommended by the standard guideline. The readings are taken at 15-minute intervals for the initial hour, hourly from the first to the sixth hour, every six hours from 6 to 24 hours, and then twice daily for 7 days (or death, if earlier). Subsequently, these data are uploaded into the research database.
  Arms: Intervention group
Other: Control group — After stroke progression, all patients receive dual antiplatelet therapy (aspirin 100mg/day combined with clopidogrel 75mg/day) for the first 21 days, except in cases of cerebral hemorrhage. After this period, they continue to take aspirin 100mg/day orally for the long term.
  Arms: Control group

SUMMARY:
Stroke has become the leading cause of death in China, with acute ischemic stroke still progressing within one week of onset, known as progressive ischemic stroke (PIS), which has a high rate of disability and mortality, accounting for 23-43% of the incidence of stroke. Non-cardioembolic PIS is one of the common types, and the current treatment mainly focuses on antithrombotic therapy, but the therapeutic effect is not satisfactory. More and more evidence suggests that hypotension is an unfavorable factor for PIS, so this study intends to explore the efficacy and safety of antithrombotic therapy with regulation of blood pressure in non-cardioembolic PIS.

DETAILED DESCRIPTION:
This is a single-center randomized controlled study conducted to explore the efficacy and safety of antithrombotic therapy with regulation of blood pressure in non-cardioembolic PIS.

We plan to recruit 70 patients with non-cardioembolic PIS. All subjects are of Han ethnicity, aged 18 years or older. Gender and age will be statistical data after enrollment. Patients will participate in the study after informed consent.

Then patients who meet the inclusion and exclusion criteria will be randomly assigned in a 1:1 ratio to the control group (antithrombotic therapy) or the intervention group (antithrombotic + blood pressure control therapy). In addition to antithrombotic therapy, the intervention group will use medications such as dopamine, metaraminol, or midodrine to control systolic blood pressure within the range of 160-180 mmHg and maintain it for one week.

Patients will be followed up at 2 weeks for mRS (Modified Rankin Scale) and NIHSS (National Institutes of Health Stroke Scale) scores，and at one month for mRS scores, and at three months for mRS and BI (Barthel Index) scores.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged ≥18 years) with an AIS who have been able to complete usual activities in daily life without support before the stroke;
2. One of the following PIS manifestations:

   1. Within 7 days of onset, when symptom worsens and there are new lesions or infarct growth on DWI within 24 hours of aggravation, the National Institutes of Health Stroke Scale (NIHSS) score increases by ≥ 2 points ;
   2. Within 24 hours after IVT, when symptom worsens and there are new lesions or infarct growth on DWI within 24 hours of aggravation, the NIHSS score increases by ≥ 4 points compared to the baseline;
3. Within 3h of stroke progression, ≥2 successive measurements of systolic blood pressure (SBP) < 160 mm Hg for >10 min.
4. Computed tomographic angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA) confirms patients without visible large or medium-sized intracranial vessel occlusion.

Exclusion Criteria:

1. After stroke progression, a head CT confirmed new cerebral hemorrhage or hemorrhagic transformation.
2. Endovascualr treatment had been performed before stroke progression (thrombectomy, stent placement, balloon dilatation) or if surgery or interventional treatment had been scheduled;
3. Current treatment with heparin therapy or oral anticoagulation (presumed cardiac source of embolus, such as atrial fibrillation, prosthetic cardiac valve, and known or suspected endocarditis);
4. Previous diseases of the brain that include intracranial hemorrhage or amyloid angiopathy; brain surgery or hemorrhagic stroke; stroke within the last three months;
5. Preexisting serious diseases: Cancer, AIDS, serious heart disease, dementia, liver diseases such as liver failure, cirrhosis, portal hypertension and active hepatitis, acute or chronic severe renal impairment (glomerular filtration rate < 30 ml/min/1·73 m2 );
6. Contraindication to aspirin or clopidogrel;
7. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with an excellent outcome（mRS score 0-1）at 90 days after randomization | at 90 days after randomization
  modified Rankin scale (mRS，an ordinal global disability scale with scores ranging from 0 [no symptoms] to 6 [death]) at 90 days after randomization. An excellent outcome is defined as score of 0 or 1 on the mRS score at 90 days.

SECONDARY OUTCOMES:
proportion of patients with outcome measured by the Barthel index (BI) | at 90 days after randomization
  outcome measured by the Barthel index (BI)，≥ 95 for the BI
proportion of patients with outcome measured by mRS | at 90 days after randomization
  outcome measured by mRS，0-2 for mRS
proportion of patients with an excellent outcome | at 2 weeks after randomization and at day 30 after randomization
  proportion of patients with an excellent outcome（0-1 for the mRS）
proportion of patients with functional independence | at 2 weeks after randomization and at day 30 after randomization
  proportion of patients with functional independence (0-2 for the mRS)
proportion of patients with outcome measured by NIHSS | at 2 weeks after randomization
  outcome measured by NIHSS (0-1 for the NIHSS)
proportion of patients with severe or moderate bleeding | at 90 days after randomization
  severe or moderate bleeding，as defined by the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) criteria
proportion of patients with any bleeding | at 90 days after randomization
  any bleeding，such as nasal bleeding, gingival bleeding, skin ecchymosis, etc.
proportion of patients with death | at 90 days after randomization
  all cause of death
proportion of patients with adverse events | at 90 days after randomization
  adverse events，such as allergic reaction，symptoms of hypertensive encephalopathy，etc.
proportion of patients with severe adverse events | at 90 days after randomization
  severe adverse events, as defined by serious drug side effects and serious unexpected events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin North Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data for the analyses
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: the study has finished
Access Criteria: contact to the primary investigator

REFERENCES:
- [Background] Helleberg BH, Ellekjaer H, Indredavik B. Outcomes after Early Neurological Deterioration and Transitory Deterioration in Acute Ischemic Stroke Patients. Cerebrovasc Dis. 2016;42(5-6):378-386. doi: 10.1159/000447130. Epub 2016 Jun 29. PMID 27351585
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Effect of blood pressure and diabetes on stroke in progression. Lancet. 1994 Jul 16;344(8916):156-9. doi: 10.1016/s0140-6736(94)92757-x. PMID 7912765
- [Background] Yang P, Song L, Zhang Y, Zhang X, Chen X, Li Y, Sun L, Wan Y, Billot L, Li Q, Ren X, Shen H, Zhang L, Li Z, Xing P, Zhang Y, Zhang P, Hua W, Shen F, Zhou Y, Tian B, Chen W, Han H, Zhang L, Xu C, Li T, Peng Y, Yue X, Chen S, Wen C, Wan S, Yin C, Wei M, Shu H, Nan G, Liu S, Liu W, Cai Y, Sui Y, Chen M, Zhou Y, Zuo Q, Dai D, Zhao R, Li Q, Huang Q, Xu Y, Deng B, Wu T, Lu J, Wang X, Parsons MW, Butcher K, Campbell B, Robinson TG, Goyal M, Dippel D, Roos Y, Majoie C, Wang L, Wang Y, Liu J, Anderson CS; ENCHANTED2/MT Investigators. Intensive blood pressure control after endovascular thrombectomy for acute ischaemic stroke (ENCHANTED2/MT): a multicentre, open-label, blinded-endpoint, randomised controlled trial. Lancet. 2022 Nov 5;400(10363):1585-1596. doi: 10.1016/S0140-6736(22)01882-7. Epub 2022 Oct 28. PMID 36341753

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT06551727/Prot_SAP_002.pdf
  • Informed Consent Form (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT06551727/ICF_001.pdf